CLINICAL TRIAL: NCT04888273
Title: Assessing the Feasibility of an Intervention for Youth and Parents Transitioning From Pediatric to Adult Eating Disorder Services: A Mixed Methods Study
Brief Title: Assessing the Feasibility of an Intervention for Youth and Parents Transitioning to Adult Eating Disorder Services
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Jennifer Couturier, Principal Investigator, McMaster University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 13303
Record Dates: First submitted 2021-04-28; First posted 2021-05-17 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Eating Disorders; Eating Disorders in Adolescence
Keywords: healthcare transition; health services; adolescent medicine
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All adolescents and parents who meet the eligibility criteria (Experimental): The adolescents and parents will be invited to participate in a 5-component intervention that will hopefully empower and prepare the pair for the transition to adult care.
  Interventions: Behavioral: Transition Intervention

INTERVENTIONS:
Behavioral: Transition Intervention — Each adolescent-parent pair will be invited to complete 5 components of the intervention (peer support session, parent education session, transition meeting with healthcare providers, family doctor contact, and reading a transition navigation guide) over a 3-month period. These intervention components were designed with the intention of making the transition process transparent for the duo, preparing the adolescent to take responsibility of their own health as it relates to their disorder, and helping the parent step back from the process to help the adolescent integrate to adult care better.

SUMMARY:
Teenagers with eating disorders often experience a disruption in care upon turning 18. At this age, they are no longer eligible to receive pediatric treatment but are also not yet set up with the appropriate adult services. There are currently no supports in place to help youth with eating disorders and their families during this transition from child to adult care. In this project, the investigators will be implementing an intervention designed to improve this transition experience; it will include peer support, parent education, a meeting with the child and adult care providers, contact with the family doctor, and a written guide about the transition. Among 10 adolescent-parent pairs leaving McMaster Children's Hospital to adult programs in Hamilton, Ontario, the investigators will assess how feasible the intervention is to implement, how feasible the chosen measures are, participants' experience of the intervention, how many adolescents actually transition to adult care, as well as a few adolescent and parent outcomes, such as how prepared the teen feels or what the parents' needs are.

DETAILED DESCRIPTION:
Eating disorders (EDs) are severe psychiatric illnesses that negatively impact the health and quality of life of sufferers and their families. EDs typically begin in adolescence and often progress into adulthood, often requiring youth to transition from pediatric to adult mental health services. However, patients often experience a discontinuity in care due to a lack of coordinated transition between services, which has a significant impact on their health. Although barriers to a smooth transition and solutions to mend the gap have been identified in the literature, there is no stakeholder-informed protocol in Canada to address this issue.

The aim of this project is to develop and test a protocol to support the health services transition from pediatric to adult treatment for adolescents with EDs and their families.

The investigators have prepared a protocol aimed at improving this transition experience using suggestions from the existing literature. The investigators will also invite stakeholders to offer recommendations for its local use. The proposed suite of interventions will be tested in a sample of adolescents who are in treatment at a pediatric ED program based in Hamilton, Ontario during their transition to adult services, along with their parents. The investigators will report upon enrolment and retention rates into adult programs, feasibility indicators of the intervention and research procedures, self-reported readiness to transition, post-transition qualitative interviews with adolescents and parents regarding their experience, and written reflections by all participants regarding each intervention component. The eligibility criteria and outcome measures will be elaborated upon below.

If this study is successful, the investigators will test the feasibility, acceptability, and cost of this protocol across pediatric ED programs in Ontario, and eventually Canada. This innovative protocol has the potential to improve health outcomes for this population, to decrease long-term disability costs associated with EDs, and to improve the quality and success of the mental health service delivery that directly influences the quality of life of Canadian youth and families affected by EDs.

ELIGIBILITY:
Inclusion Criteria for Adolescents:

* 3-6 months away from 18th birthday
* Be currently diagnosed with an ED
* Enrolled at McMaster Children's Hospital's Pediatric Eating Disorder Program
* Be in the process of preparing for a healthcare transition to local adult ED services based on pediatric healthcare providers' recommendation

Inclusion Criteria for Parents:

* Must be the parent of an adolescent who meets the criteria above

Inclusion Criteria for Adolescents and Parents

* English-speaking
* Access to a working computer with a functioning microphone and regular internet connection

Ages: 17 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Proportion of Intervention Components Completed | Post-Intervention (12 weeks)
  The investigators will capture the proportion of intervention components that were completed. This outcome will help to gather an understanding of the feasibility of the intervention. This quantitative outcome will be collected through Qualtrics via the Reflection Entries; these are short qualitative journal entries with prompts that each participant is asked to complete after completing each intervention component throughout their 3-month intervention period. The results regarding this outcome will be reported in a descriptive summary at the end of the study and integrated with the other data related to the feasibility of the intervention, both qualitative and quantitative.
Type of Intervention Components Completed | Post-Intervention (12 weeks)
  The investigators will capture which of intervention components were completed as a feasibility indicator of the intervention. This outcome will help to gather an understanding of the feasibility of the intervention. This quantitative outcome will be collected through Qualtrics via the Reflection Entries. The results regarding this outcome will be reported in a descriptive summary at the end of the study and integrated with the other data related to the feasibility of the intervention, both qualitative and quantitative.
Average Duration of Time to Complete Each Intervention Component | Post-Intervention (12 weeks)
  The investigators will capture how much time it took to complete each intervention components as a feasibility indicator of the intervention. This outcome will help to gather an understanding of the feasibility of the intervention. This quantitative outcome will be collected through Qualtrics via the Reflection Entries. The results regarding this outcome will be reported in a descriptive summary at the end of the study and integrated with the other data related to the feasibility of the intervention, both qualitative and quantitative.
Average Duration of Time to Complete the Intervention | Post-Intervention (12 weeks)
  The investigators will capture how much time it took to complete the entire intervention as a feasibility indicator of the intervention. This outcome will help to gather an understanding of the feasibility of the intervention. This quantitative outcome will be collected through Qualtrics via the Reflection Entries. The results regarding this outcome will be reported in a descriptive summary at the end of the study and integrated with the other data related to the feasibility of the intervention, both qualitative and quantitative.
Adolescent Perceptions of the Feasibility of the Intervention | Post-Intervention (12 weeks)
  The investigators will capture adolescent perceptions of feasibility of the entire intervention in the Post-Intervention Adolescent Interview. The quantitative and qualitative data related to this primary mixed methods outcome (Feasibility of the Intervention) will be integrated together at the data analysis phase.
Parent Perceptions of the Feasibility of the Intervention | Post-Intervention (12 weeks)
  The investigators will capture parent perceptions of feasibility of the entire intervention in the Post-Intervention Parent Interview. The quantitative and qualitative data related to this primary mixed methods outcome (Feasibility of the Intervention) will be integrated together at the data analysis phase.
Adolescent Perceptions of the Feasibility of the Each Intervention Component | Throughout the participant's intervention period (0 to 12 weeks)
  The investigators will capture adolescent perceptions of feasibility of the entire intervention in the Reflection Entries. The quantitative and qualitative data related to this primary mixed methods outcome (Feasibility of the Intervention) will be integrated together at the data analysis phase.
Parent Perceptions of the Feasibility of the Each Intervention Component | Throughout the participant's intervention period (0 to 12 weeks)
  The investigators will capture parent perceptions of feasibility of the entire intervention in the Reflection Entries. The quantitative and qualitative data related to this primary mixed methods outcome (Feasibility of the Intervention) will be integrated together at the data analysis phase.

SECONDARY OUTCOMES:
Study Interest Rate | 10 months after baseline
  The investigators will calculate the interest rate of the study: the numerator will be the number of adolescent-parent dyads who complete the Contact Information Form or reach out to the investigator about the study and the denominator will be the number of eligible dyads during the study period at the study site. This quantitative outcome will help to gather an understanding of the feasibility of the research procedures and methods of the study and will be collected through Qualtrics via the Reflection Entries. The results regarding this outcome will be reported in a descriptive summary at the end of the study and integrated with the other data related to the feasibility of the research procedures and methods, both qualitative and quantitative.
Study Recruitment Rate | 10 months after baseline
  The investigators will calculate the recruitment rate of the study: the numerator will be the number of dyads that are enrolled in the study (i.e., signed consent) and the denominator will be the number of adolescent-parent dyads who complete the Contact Information Form or reach out to the investigator about the study. This quantitative outcome will help to gather an understanding of the feasibility of the research procedures and methods of the study and will be collected through Qualtrics via the Reflection Entries. The results regarding this outcome will be reported in a descriptive summary at the end of the study and integrated with the other data related to the feasibility of the research procedures and methods, both qualitative and quantitative.
Study Completion Rate | 10 months after baseline
  The investigators will calculate the completion rate of the study: the numerator will be the number of dyads that complete the study (i.e., post-intervention measures) and the denominator will be the number of dyads that are enrolled in the study (i.e., signed consent). This quantitative outcome will help to gather an understanding of the feasibility of the research procedures and methods of the study and will be collected through Qualtrics via the Reflection Entries. The results regarding this outcome will be reported in a descriptive summary at the end of the study and integrated with the other data related to the feasibility of the research procedures and methods, both qualitative and quantitative.
Proportion of Missing Data | 10 months after baseline
  The investigators will calculate the proportion of missing data (i.e., individual questions, entire surveys) across all data collection measures. This quantitative outcome will help to gather an understanding of the feasibility of the research procedures and methods of the study. The results regarding this outcome will be reported in a descriptive summary at the end of the study and integrated with the qualitative data regarding this outcome at the data analysis stage.
Average Duration of Time to Complete Data Collection Measures | 10 months after baseline
  The investigators will calculate the duration of time it takes participants to complete each data collection measure (i.e., individual surveys, interviews). This quantitative outcome will help to gather an understanding of the feasibility of the research procedures and methods of the study. The results regarding this outcome will be reported in a descriptive summary at the end of the study and integrated with the qualitative data regarding this outcome at the data analysis stage.
Adolescent Perceptions of the Feasibility of the Research Procedures and Methods | Post-Intervention (12 weeks)
  The investigators will capture adolescent perceptions of the feasibility of the research procedures and the methods using the Post-Intervention Adolescent Interview (specifically, perceptions of response burden and measure relevance). The quantitative and qualitative data related to this secondary mixed methods outcome (Feasibility of the Research Procedures and Methods) will be integrated together at the data analysis phase.
Parent Perceptions of the Feasibility of the Research Procedures and Methods | Post-Intervention (12 weeks)
  The investigators will capture parent perceptions of the feasibility of the research procedures and the methods using the Post-Intervention Parent Interview (specifically, perceptions of response burden and measure relevance). The quantitative and qualitative data related to this secondary mixed methods outcome (Feasibility of the Research Procedures and Methods) will be integrated together at the data analysis phase.
Adolescent Experience of the Intervention | Throughout the participant's intervention period (0 to 12 weeks) and at Post-Intervention (12 weeks)
  The investigators will capture the experience of the intervention from the adolescent using the Reflection Entries and the Post-Intervention Adolescent Interview. Specifically, this will include asking about their self-reported experience, preferences for the components, and feedback about the intervention.
Parent Experience of the Intervention | Throughout the participant's intervention period (0 to 12 weeks) and at Post-Intervention (12 weeks)
  The investigators will capture the experience of the intervention from the parent using the Reflection Entries and the Post-Intervention Parent Interview. Specifically, this will include asking about their self-reported experience, preferences for the components, and feedback about the intervention.
Enrolment and Retention to Adult Care | 1 month after the participating adolescent's 18th birthday
  The investigators will re-contact the adolescents in the study to capture the proportion of adolescents that transitioned to adult care to see if they enrolled and are continuing to attend adult care. This quantitative outcome will be reported as a proportion.
Change in Adolescent's Range and Severity of Eating Disorder Symptoms - Eating Disorder Examination Questionnaire | At Baseline (0 weeks) and Post-Intervention (12 weeks) of each adolescent's time in the intervention
  The investigators will capture the adolescent's self-reported range and severity of their eating disorder symptoms before and after the adolescent completes the intervention using the Eating Disorder Examination Questionnaire (EDE-Q 6.0). This measure contains 22 Likert-scale items (from 0 to 6). The minimum total score for these questions is 0 and the maximum is 132. Higher scores indicate an increased range and/or severity of eating disorder symptoms. The measure also contains 6 self-report questions where respondents are asked to report the frequency of a behaviour (e.g., restricting) and their height, weight, and menstrual patterns (if applicable).
  Repeated Measures design will be used to analyze the mean difference in total score of this measure from baseline to post-intervention. A descriptive summary of the responses to the differently-formatted questions (items related to behaviour frequency, height, weight, and menstrual patterns) will be reported as well.
Change in Adolescent's Level of Readiness for Transition - Transition Readiness Assessment Questionnaire | At Baseline (0 weeks) and Post-Intervention (12 weeks) of each adolescent's time in the intervention
  The investigators will capture the adolescent's self-reported level of readiness for transition to adult care before and after the adolescent completes the intervention using the Transition Readiness Assessment Questionnaire (TRAQ). This skill-focused tool contains 20 Likert-scale questions (from 1 to 5 in increments of 1) organized by 5 domains: medication management, appointment management, health issue tracking, interactions with providers, and daily activity management. The minimum total score of this tool is 20 and the maximum total score is 100. Higher scores indicate increased readiness for transition.
  Repeated Measures design will be used to analyze the mean difference in total score of this measure from baseline to post-intervention.
Change in Adolescent's Awareness of their Eating Disorder and Ability to Make Healthcare-Relevant Decisions - Self-Management Skills Assessment Guide (Youth Report) | At Baseline (0 weeks) and Post-Intervention (12 weeks) of each adolescent's time in the intervention
  The investigators will capture the adolescent's self-reported awareness of their health condition and ability to make decisions relevant to their healthcare needs before and after the adolescent completes the intervention using the Self-Management Skills Assessment Guide (Youth Report) (SMSAG-Y). This measure contains 21-identically structured Likert-scale items (from 1 to 5 in increments of 1). The minimum total score of this tool is 21 and the maximum total score is 105. Higher scores indicate increased awareness and ability surrounding their eating disorder.
  Repeated Measures design will be used to analyze the mean difference in total score of this measure from baseline to post-intervention. Additionally, since this measure will also be completed by the parent, the scores will compared to assess similarities and differences between their perspectives.
Change in Adolescent's Readiness and Motivation to Change Eating Disorder Symptoms and Behaviours - Eating Disorders Readiness Ruler | At Baseline (0 weeks) and Post-Intervention (12 weeks) of each adolescent's time in the intervention
  The investigators will capture the adolescent's self-reported readiness and motivation to change various eating disorder behaviours before and after the adolescent completes the intervention using the Eating Disorders Readiness Ruler (ED-RR). The first 9 items (from 1 to 10) measure readiness to change (minimum score of 9 to a maximum of 90). Higher scores for these items indicates increased willingness to change. The last 9 items measure the extent to which the change is being made for others versus for themselves on a scale from 10% to 100%. A "controlled motivation" score of 1 is assigned to responses from 0 to 30% (change is for others) and an "autonomous motivation" score of 1 is assigned to responses from 80-100% (change is for themselves). Total scores for each motivation type are computed, ranging from 0 to 9.
  Repeated Measures design will be used to analyze the mean difference in the total score for each domain from baseline to post-intervention.
Change in Parent's Perceived Burden and Impact of Child's Eating Disorder Symptoms on Their Lives - Eating Disorder Symptom Impact Scale | At Baseline (0 weeks) and Post-Intervention (12 weeks) of each parent's time in the intervention
  The investigators will capture the parent's self-reported carer burden and impact of eating disorder symptoms on parents' lives before and after the parent completes the intervention using the Eating Disorders Symptom Impact Scale (EDSIS). This measure has 24 Likert-scale items (from 0 to 4 in increments of 1) on four domains: nutrition, guilt, unregulated behaviour, and social isolation. The minimum total score of this measure is 0 and the maximum total score is 96. Higher scores indicate increased burden or impact of their child's disorder on the respondent.
  Repeated Measures design will be used to analyze the mean difference in total score of this measure from baseline to post-intervention.
Change in Parent's Perceived Needs as a Carer of an Individual with an Eating Disorder- Carers Needs Assessment Measure | At Baseline (0 weeks) and Post-Intervention (12 weeks) of each parent's time in the intervention
  The investigators will capture the parent's self-reported needs as the carer of an individual with an eating disorder before and after the parent completes the intervention using the Carers Needs Assessment Measure (CaNAM). This tool contains 32 Likert-scale items (from 0 to 2) across three domains: information about eating disorders, support from people/organizations, and support for yourself (minimum total score of 0 and maximum of 64). Higher scores indicate that the respondent is satisfied with the resources/information they've received. The final domain contains 15 yes/no questions regarding areas where the respondent may appreciate help. The 4 remaining open-ended questions ask the respondent elaborate upon each domain.
  Repeated Measures design will be used to analyze the mean difference in total score and subscales of this measure from baseline to post-intervention. A descriptive summary will be used to summarize the responses to the open-ended questions.
Change in Parent Self-Efficacy and Collaboration with Other Parents - Patient and Carer Collaboration Scale | At Baseline (0 weeks) and Post-Intervention (12 weeks) of each parent's time in the intervention
  The investigators will capture the parent's self-reported self-efficacy and collaboration among carers of patients with an eating disorder before and after the parent completes the intervention using the Patient and Carer Collaboration Scale - Carer (PACCS-C). This measure is comprised of 33 Likert-scale questions (from 0 to 100 in increments of 10) that relate to four constructs: hope, self-care and compassion, externalization of the eating disorder, and boundaries. The minimum total score of this measure is 0 and the maximum total score is 3300. Higher scores indicate better outcomes (e.g., setting strong boundaries, increased hope).
  Repeated Measures design will be used to analyze the mean difference in total score and subscales of this measure from baseline to post-intervention.
Change in Parent's Perception of their Child's Awareness of their Eating Disorder and Ability to Make Healthcare-Relevant Decisions - Self-Management Skills Assessment Guide (Parent Report) | At Baseline (0 weeks) and Post-Intervention (12 weeks) of each parent's time in the intervention
  The investigators will capture the parent's self-reported perception of their child's awareness of their health condition and the child's ability to make healthcare decisions before and after the parent completes the intervention using the Self-Management Skills Assessment Guide (Parent Report) (SMSAG-P). This measure contains 22-identically structured Likert-scale items (from 1 to 3 in increments of 1) where higher scores indicate the parent's increased belief in their child's awareness and ability surrounding their eating disorder. The minimum total score of this tool is 22 and the maximum total score is 66.
  Repeated Measures design will be used to analyze the mean difference in total score of this measure from baseline to post-intervention. Additionally, since this measure will also be completed by the adolescent, the scores will compared to assess similarities and differences between their perspectives.
Adolescent Demographics | At Baseline (0 weeks) of each adolescent's time in the intervention
  In the baseline measure package, that includes the adolescent outcome measures above, the investigators will ask the adolescent their sex, gender, date of birth, school grade, ethnicity, type of eating disorder, length of eating disorder, date of diagnosis, and type of treatment received to date. A descriptive summary of demographic information will be prepared to report this data.
Parent Demographics | At Baseline (0 weeks) of each parent's time in the intervention
  In the baseline measure package, that includes the parent outcome measures above, the investigators will ask the parent their sex, gender, age, ethnicity, relationship to adolescent (e.g., parent, stepparent, guardian), marital status, household income, highest level of education achieved, number of people in household, number of children cared for, number of children (apart from participating adolescent) who have an eating disorder and corresponding details, and whether the parent has had an eating disorder and corresponding details. A descriptive summary of demographic information will be prepared to report this data.

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster Children's Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nicula M, Kimber M, Boylan K, Grant C, Laliberte M, Miller K, Dimitropoulos G, Trollope K, Webb C, Couturier J. Assessing the feasibility of an intervention for adolescents and parents transitioning out of paediatric eating disorder services: A mixed methods study. Eur Eat Disord Rev. 2025 Nov;33(6):1144-1161. doi: 10.1002/erv.3027. Epub 2023 Aug 26. PMID 37632341